CLINICAL TRIAL: NCT03711279
Title: A Multicenter, Randomized, Open, Phase 2 Trial of SHR-1210 Plus Apatinib Versus Doxorubicin (ADM) Plus Ifosfamide (IFO) in Patients With Soft Tissue Sarcoma
Brief Title: A Study of SHR-1210 Plus Apatinib in Patients With Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor R & D Strategy Adjustment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II-212
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2023-07

CONDITIONS: Sarcoma
Keywords: Sarcoma; SHR-1210; Apatinib
MeSH Terms: conditions — Sarcoma | interventions — camrelizumab; apatinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1210 plus Apatinib (Experimental)
  Interventions: Drug: SHR-1210 plus Apatinib
- ADM plus IFO or IFO alone (Active Comparator)
  Interventions: Drug: ADM plus IFO or IFO alone

INTERVENTIONS:
Drug: SHR-1210 plus Apatinib — SHR-1210 200 mg q3w+ Apatinib 500 mg qd
  Other Names: PD-1 antibody + Anti-angiogenesis
  Arms: SHR-1210 plus Apatinib
Drug: ADM plus IFO or IFO alone — ADM 60 mg/m2 D1 + IFO 2 g/m2 D1-D4 q3w；if the cumulative doses of ADM were beyond 450 mg/m2, the monotherapy of IFO (2 g/m2 D1-D5 q3w) would be used.
  Other Names: chemotherapy
  Arms: ADM plus IFO or IFO alone

SUMMARY:
The main purpose of this study is to evaluate the efficacy of SHR-1210 plus Apatinib versus AMD plus IFO in participants with soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with the age from 16 years to 70 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;the ECOG performance status of 2 can be accepted after the amputation.
* Life expectancy of at least 3 months.
* Histologically confirmed diagnosis of advanced unresectable or metastatic soft tissue sarcoma not amenable to curative treatment with surgery or radiotherapy.The histopathologic types as specified in the protocol.
* Without prior systemic chemotherapy or relapse more than 6 months after the completion of last systemic chemotherapy.
* Presence of measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Acceptable liver function, renal function, hematologic status and coagulation function as specified in the protocol.
* Females of child-bearing potential must have a negative serum pregnancy test within 7 days prior to randomization.Females of child-bearing potential and males must agree to use highly effective contraceptive precautions during the trial and up to 3 months following the last dose of study drug.
* Willingness to comply with the study protocol for any reason.

Exclusion Criteria:

* Receiving any previous anticancer treatment, other investigational drugs or any attenuated live vaccine with 4 weeks of the first does of study drug.
* Prior treatment with PD-1/PD-L1/CTLA-4 targeted drugs or VEGFR targeted drugs.
* Plan to receive surgery or radiotherapy to treat the sarcoma during the trail.
* Radiological evidence of brain metastases or primary tumors.
* Diagnosed other malignancies within the last 3 years from the first dose of drug.
* Known allergy to any of the treatment components.
* Active infection including human immunodeficiency virus (HIV) ,HBV or HCV.
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yao, M.D., Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (1):
- Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SHR-1210 Plus Apatinib | ADM Plus IFO or IFO Alone
Started | 51 | 48
Completed | 50 | 47
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SHR-1210 Plus Apatinib | ADM Plus IFO or IFO Alone | Total
Number analyzed (Participants) | 50 | 47 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 49 | 41 | 90
  >=65 years | 1 | 5 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 30 | 27 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 50 | 47 | 97
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 50 | 47 | 97

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Randomization to Radiographic Progression or Death Due to Any Cause (Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions)
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 31 months, CT was conducted at baseline、weeks 7、13、19 and then every 12 weeks.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SHR-1210 Plus Apatinib | ADM Plus IFO or IFO Alone
Number analyzed (Participants) | 50 | 47
months | 5.6 [4.1 to 6.9] | 5.5 [3.5 to 8.4]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Baseline to documented disease Remission to study discontinuation, Partial Remission is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 30% decrease in the sum of the beaseline diameter of target lesions.
Time Frame: From date of randomization until the date of study completion, an average of 1 year, CT was conducted at baseline、weeks 7、13、19 and then every 12 weeks.
Measure: Number; unit: participants
Arm/Group | SHR-1210 Plus Apatinib | ADM Plus IFO or IFO Alone
Number analyzed (Participants) | 50 | 47
participants | 11 | 5

ADVERSE EVENTS:
Time Frame: 18 months
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | SHR-1210 Plus Apatinib | ADM Plus IFO or IFO Alone
All-Cause Mortality (participants affected / at risk) | 2/50 | 2/47
Serious Adverse Events (participants affected / at risk) | 27/50 | 13/47
Other Adverse Events (participants affected / at risk) | 50/50 | 45/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SHR-1210 Plus Apatinib (N=50) | ADM Plus IFO or IFO Alone (N=47)
Drug-induced liver injury (Hepatobiliary disorders) | 3 | 0
Liver injury (Hepatobiliary disorders) | 2 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 5
Lymphocyte count decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 0 | 4
Neutrophil count decreased (Investigations) | 0 | 5
Pyrexia (General disorders) | 3 | 1
Impaired healing (General disorders) | 1 | 0
Hernia (General disorders) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Cor Pulmonale (Cardiac disorders) | 1 | 0
Degenerative aortic valve disease (Cardiac disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Myelosuppression (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SHR-1210 Plus Apatinib (N=50) | ADM Plus IFO or IFO Alone (N=47)
Anaemia (Blood and lymphatic system disorders) | 21 | 34
Coagulopathy (Blood and lymphatic system disorders) | 3 | 0
Sinus tachycardia (Cardiac disorders) | 8 | 0
Hypothyroidism (Endocrine disorders) | 20 | 1
Hyperthyroidism (Endocrine disorders) | 8 | 0
Diarrhoea (Gastrointestinal disorders) | 25 | 3
Mouth ulceration (Gastrointestinal disorders) | 18 | 4
Nausea (Gastrointestinal disorders) | 17 | 23
Vomiting (Gastrointestinal disorders) | 17 | 20
Constipation (Gastrointestinal disorders) | 16 | 17
Abdominal pain upper (Gastrointestinal disorders) | 7 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Stomatitis (Gastrointestinal disorders) | 5 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 2
Abdominal pain lower (Gastrointestinal disorders) | 3 | 2
Gingival pain (Gastrointestinal disorders) | 3 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 15 | 12
Pyrexia (General disorders) | 15 | 6
Chest discomfort (General disorders) | 7 | 4
Chest pain (General disorders) | 4 | 1
Fatigue (General disorders) | 3 | 1
Oedema peripheral (General disorders) | 3 | 0
Reactive capillary endothelial proliferation (Immune system disorders) | 8 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 2
Urinary tract infection (Infections and infestations) | 7 | 4
Nasopharyngitis (Infections and infestations) | 6 | 1
Pneumonia (Infections and infestations) | 4 | 2
Aspartate aminotransferase increased (Investigations) | 33 | 9
Alanine aminotransferase increased (Investigations) | 31 | 16
White blood cell count decreased (Investigations) | 28 | 24
Platelet count decreased (Investigations) | 26 | 18
Gamma-glutamyltransferase increased (Investigations) | 25 | 8
Weight decreased (Investigations) | 23 | 6
Neutrophil count decreased (Investigations) | 21 | 20
Blood alkaline phosphatase increased (Investigations) | 20 | 5
Blood bilirubin increased (Investigations) | 20 | 3
Lymphocyte count decreased (Investigations) | 19 | 26
Blood thyroid stimulating hormone increased (Investigations) | 15 | 0
Blood lactate dehydrogenase increased (Investigations) | 14 | 4
Bilirubin conjugated increased (Investigations) | 13 | 2
Blood bilirubin unconjugated increased (Investigations) | 10 | 1
Electrocardiogram T wave abnormal (Investigations) | 8 | 4
Total bile acids increased (Investigations) | 7 | 2
Blood albumin decreased (Investigations) | 6 | 6
Red blood cells urine positive (Investigations) | 5 | 1
Blood creatine phosphokinase MB increased (Investigations) | 4 | 0
Blood creatine phosphokinase increased (Investigations) | 4 | 0
Blood pressure increased (Investigations) | 4 | 0
Blood uric acid increased (Investigations) | 4 | 0
Fibrin D dimer increased (Investigations) | 4 | 0
Occult blood positive (Investigations) | 4 | 0
Urinary occult blood positive (Investigations) | 4 | 2
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 3 | 1
Blood creatinine increased (Investigations) | 3 | 3
Blood fibrinogen increased (Investigations) | 3 | 1
C-reactive protein increased (Investigations) | 3 | 1
Interleukin level increased (Investigations) | 3 | 0
Mitochondrial aspartate aminotransferase increased (Investigations) | 3 | 2
Neutrophil count increased (Investigations) | 3 | 3
Tri-iodothyronine free decreased (Investigations) | 3 | 0
White blood cell count increased (Investigations) | 3 | 3
Protein urine present (Investigations) | 1 | 3
Red blood cell count decreased (Investigations) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 16 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 12 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 3 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Headache (Nervous system disorders) | 16 | 4
Dizziness (Nervous system disorders) | 10 | 5
Insomnia (Psychiatric disorders) | 4 | 2
Proteinuria (Renal and urinary disorders) | 29 | 3
Haematuria (Renal and urinary disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 23 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 21 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 21
Blister (Skin and subcutaneous tissue disorders) | 3 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 3
Hypertension (Vascular disorders) | 29 | 1
Hypotension (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT03711279/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT03711279/SAP_001.pdf